CLINICAL TRIAL: NCT04759131
Title: A Phase 3 Open-label, Multicenter Study of the Safety, Efficacy, and Pharmacokinetics of Intravenous Recombinant Coagulation Factor VIII Fc-von Willebrand Factor-XTEN Fusion Protein (rFVIIIFc-VWF-XTEN; BIVV001) in Previously Treated Pediatric Patients <12 Years of Age With Severe Hemophilia A
Brief Title: Safety, Efficacy and PK of BIVV001 in Pediatric Patients With Hemophilia A
Acronym: XTEND-Kids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC16295; 2020-000769-18 (EudraCT Number); U1111-1244-0558 (Other: UTN); 017464 (Other: IND)
Record Dates: First submitted 2021-02-13; First posted 2021-02-18 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BIVV001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIVV001: Participants aged <6 Years (Experimental): Participants aged less than (<) 6 years received BIVV001 at a dose of 50 international units per kilogram (IU/kg) intravenous (IV) injection once-weekly (QW) prophylaxis for 52 weeks.
  Interventions: Drug: efanesoctocog alfa (BIVV001)
- BIVV001: Participants aged 6 to <12 Years (Experimental): Participants aged 6 to <12 years received BIVV001 at a dose of 50 IU/kg IV injection QW prophylaxis for 52 weeks.
  Interventions: Drug: efanesoctocog alfa (BIVV001)

INTERVENTIONS:
Drug: efanesoctocog alfa (BIVV001) — Pharmaceutical form: solution for injection Route of administration: IV

SUMMARY:
Primary Objective:

- To evaluate the safety of BIVV001 in previously treated pediatric participants with hemophilia A.

Secondary Objectives:

* To evaluate the efficacy of BIVV001 as a prophylaxis treatment.
* To evaluate the efficacy of BIVV001 in the treatment of bleeding episodes.
* To evaluate BIVV001 consumption for prevention and treatment of bleeding episodes.
* To evaluate the effect of BIVV001 prophylaxis on joint health outcomes.
* To evaluate the effect of BIVV001 prophylaxis on Quality of Life (QoL) outcomes.
* To evaluate the efficacy of BIVV001 for perioperative management.
* To evaluate the safety and tolerability of BIVV001 treatment.
* To assess the pharmacokinetics (PK) of BIVV001.

DETAILED DESCRIPTION:
Study duration per participants was approximately 60 weeks (maximum 8 weeks for screening and 52 weeks of treatment).

All participants completing or remaining at the end of study were offered participation in the planned extension trial.

ELIGIBILITY:
Inclusion criteria :

* Participant must be younger than 12 years of age, at the time of signing the informed consent.
* Severe hemophilia A defined as <1 international units per deciliter (IU/dL) (<1 percent [%]) endogenous Factor VIII (FVIII) as documented either by central laboratory testing at Screening or in historical medical records from a clinical laboratory demonstrating <1% FVIII coagulant activity (FVIII:C) or a documented genotype known to produce severe hemophilia A.
* Previous treatment for hemophilia A (prophylaxis or on-demand) with any recombinant and/or plasma-derived FVIII, or cryoprecipitate for at least 150 exposure days (EDs) for participants aged 6 to <12 years and above 50 EDs for participants aged <6 years.
* Weight above or equal to 10 kg.

Exclusion criteria:

* History of hypersensitivity or anaphylaxis associated with any FVIII product.
* History of a positive inhibitor (to FVIII) test defined as greater than or equal to (>=) 0.6 Bethesda units (BU/mL), or any value greater than or equal to the lower sensitivity cut-off for laboratories with cut-offs for inhibitor detection between 0.7 and 1.0 BU/mL, or clinical signs or symptoms of decreased response to FVIII administrations. Family history of inhibitors would not exclude the participant.
* Positive inhibitor test result, defined as >=0.6 BU/mL at Screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Max Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (40):
- United States (10):
  - Children's Hospital Los Angeles-Site Number:8400006, Los Angeles, California
  - University of Florida-Site Number:8400009, Gainesville, Florida
  - Children's Healthcare of Atlanta-Site Number:8400019, Atlanta, Georgia
  - Rush University Medical Center-Site Number:8400001, Chicago, Illinois
  - University of Iowa Hospitals and Clinics-Site Number:8400002, Iowa City, Iowa
  - NY Presbyterian - Weill Cornell Medical Center-Site Number:8400020, New York, New York
  - East Carolina University/Brody Medical Sciences Building-Site Number:8400015, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center-Site Number:8400008, Cincinnati, Ohio
  - Childrens Hospital Of Columbus-Site Number:8400012, Columbus, Ohio
  - Children's Hospital Of Wisconsin-Site Number:8400005, Milwaukee, Wisconsin
- Australia (2):
  - Investigational Site Number :0360001, Westmead, New South Wales
  - Investigational Site Number :0360002, South Brisbane, Queensland
- Canada (4):
  - Investigational Site Number :1240004, Hamilton, Ontario
  - Investigational Site Number :1240003, London, Ontario
  - Investigational Site Number :1240002, Ottawa, Ontario
  - Investigational Site Number :1240001, Toronto, Ontario
- France (3):
  - Investigational Site Number :2500004, Bron
  - Investigational Site Number :2500001, Le Kremlin-Bicêtre
  - Investigational Site Number :2500003, Lille
- Germany (2):
  - Investigational Site Number :2760001, Frankfurt am Main
  - Investigational Site Number :2760002, München
- Investigational Site Number :3480005, Pécs, Hungary
- Investigational Site Number :3720001, Dublin, Ireland
- Italy (2):
  - Investigational Site Number :3800001, Milan
  - Investigational Site Number :3800002, Napoli
- Netherlands (2):
  - Investigational Site Number :5280002, Amsterdam
  - Investigational Site Number :5280001, Utrecht
- Spain (2):
  - Investigational Site Number :7240002, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number :7240001, Madrid, Madrid, Comunidad de
- Investigational Site Number :7520001, Malmo, Sweden
- Investigational Site Number :7560001, Zurich, Switzerland
- Taiwan (4):
  - Investigational Site Number :1580001, Taichung
  - Investigational Site Number :1580003, Taichung
  - Investigational Site Number :1580002, Taipei
  - Investigational Site Number :1580004, Taipei
- Turkey (Türkiye) (3):
  - Investigational Site Number :7920004, Antalya
  - Investigational Site Number :7920001, Istanbul
  - Investigational Site Number :7920003, Izmir
- United Kingdom (2):
  - Investigational Site Number :8260003, Birmingham
  - Investigational Site Number :8260001, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Malec L, Mathias M, Dunn AL, Nolan B, Wong N, Bystricka L, Khan U, Neill G, Santagostino E, Gunawardena S, Tarango C, Peyvandi F. Post hoc analysis of bleeding episodes and clinically relevant pharmacokinetic parameters among children <12 years old with severe hemophilia A receiving once-weekly efanesoctocog alfa prophylaxis in the XTEND-Kids phase 3 multinational trial. J Thromb Haemost. 2025 Nov;23(11):3481-3491. doi: 10.1016/j.jtha.2025.07.011. Epub 2025 Jul 21. PMID 40701256
- [Derived] Klamroth R, von Drygalski A, Hermans C, Park YS, Chan AKC, Kupesiz A, Alvarez-Roman MT, Malec L, Santagostino E, Neill G, Bystricka L, Dumont J, Abad-Franch L, Fetita LS, Khoo L. Perioperative Management With Efanesoctocog Alfa in Patients With Haemophilia A in the Phase 3 XTEND-1 and XTEND-Kids Studies. Haemophilia. 2025 May;31(3):391-400. doi: 10.1111/hae.70017. Epub 2025 Mar 18. PMID 40099428
- [Derived] Malec L, Peyvandi F, Chan AKC, Konigs C, Zulfikar B, Yuan H, Simpson M, Alvarez Roman MT, Carcao M, Staber JM, Dunn AL, Chou SC, d'Oiron R, Albisetti M, Demissie M, Santagostino E, Yarramaneni A, Wong N, Abad-Franch L, Gunawardena S, Fijnvandraat K; XTEND-Kids Trial Group. Efanesoctocog Alfa Prophylaxis for Children with Severe Hemophilia A. N Engl J Med. 2024 Jul 18;391(3):235-246. doi: 10.1056/NEJMoa2312611. PMID 39018533
- See also: EFC16295 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25243&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 40 active sites in 15 countries. A total of 79 pediatric participants were screened between 19 February 2021 to 09 February 2022, of which 5 participants had screen failure due to not meeting the eligibility criteria.
Pre-assignment Details: The study comprised of 2 age cohorts of children with severe hemophilia A: less than (<) 6 years and 6 to <12 years. A total of 74 participants were enrolled in this study.
Groups:
- BIVV001: Participants Aged <6 Years: Participants aged <6 years received BIVV001 at a dose of 50 international units per kilogram (IU/kg) intravenous (IV) injection once-weekly (QW) prophylaxis for 52 weeks.
Period: Overall Study
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Started | 38 | 36
Completed | 36 | 36
Not Completed | 2 | 0
Not completed — Investigator's discretion | 1 | 0
Not completed — Subject withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set (FAS) which included all participants who took at least 1 dose of study intervention.
Groups:
- BIVV001: Participants Aged <6 Years: Participants aged <6 years received BIVV001 at a dose of 50 IU/kg IV injection QW prophylaxis for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.69 (1.21) | 8.42 (2.08) | 5.99 (2.91)
Age, Customized [Count of Participants; unit: Participants]
  Children (1 to 5 years) | 38 | 0 | 38
  Children (>=6 to 11 years) | 0 | 36 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 36 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 4 | 8
  Race: Black or African American | 1 | 2 | 3
  Race: White | 30 | 25 | 55
  Race: Other or Not Reported | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Neutralising Antibodies (Development of Inhibitors) Directed Against Factor VIII
Description: Inhibitor development was defined as an inhibitor result of greater than or equal to (>=0.6) Bethesda units (BU/mL) that was confirmed by a second test result from a separate sample, drawn 2 to 4 weeks following the date when the original sample was drawn. Both tests must have been performed by the central laboratory using the Nijmegen modified Bethesda assay.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on safety analysis set which included all participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Participants | 0 | 0

2. Secondary Outcome: Annualized Bleeding Rate (ABR): For Treated Bleeds
Description: ABR: annualized number of treated bleeding episodes (BE) per participant per year. ABR=number of treated BE during efficacy period (EP)/total number of days during EP*365.25. Treated BE:any occurrence of hemorrhage required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat BE, any subsequent bleeding at same location/injections administered less than or equal to (<=) 72 hours apart from previous injection were considered same BE. Any injection after >72 hours post preceding one=considered 1st injection to treat new BE in same location. Any bleed at different location:considered as separate BE, regardless of time from last injection. EP=sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. ABR:by negative binomial model with total number of treated BE during EP as response variable and log transformed EP duration (years) as offset variable.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
episodes per participant per year | 0.48 [0.30 to 0.77] | 1.33 [0.64 to 2.76]

3. Secondary Outcome: Sensitivity Analysis: Annualized Bleeding Rate: For Treated Bleeds
Description: ABR: annualized number of treated BE per participant per year. ABR = number of treated BE during EP/total number of days during EP*365.25. Treated BE: any occurrence of hemorrhage that required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat BE, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same BE. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new bleeding episode in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection. EP reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. ABR: using negative binomial (NB) model with total number of treated BE during EP as response variable and log-transformed EP duration (years) as offset variable.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population. Sensitivity analysis excluded 1 participant who did not receive weekly prophylaxis treatment as specified in the protocol for an extended period of time.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
episodes per participant per year | 0.48 [0.30 to 0.77] | 0.75 [0.41 to 1.40]

4. Secondary Outcome: Annualized Bleeding Rate for All Bleeding Episodes
Description: ABR:annualized number of all BE (treated and untreated)/participant/year. ABR=number of all BE during EP/total number of days during EP*365.25. BE:any occurrence of hemorrhage required administration of BIVV001. It started from 1st sign of bleed and ended no more than 72 hours after last injection to treat BE, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same BE. Any injection after >72 hours post preceding one=considered 1st injection to treat new BE in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection. EP:sum of all intervals of time during which participants treated with BIVV001 according to study arms & treatment regimens. ABR:NB model with total number of treated BE during EP as response variable and log-transformed EP duration (years) as offset variable. Spontaneous:bleeding without contributing factor, Traumatic:bleeding with known reason.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
episodes per participant per year | 2.78 [1.39 to 5.58] | 2.85 [1.59 to 5.12]

5. Secondary Outcome: Sensitivity Analysis: Annualized Bleeding Rate for All Bleeding Episodes
Description: ABR: annualized number of all BE (treated & untreated)/participant/year. ABR=number of all BE during EP/total number of days during EP*365.25. BE: any hemorrhage occurrence required administration of BIVV001. It started from 1st sign of bleed & ended no more than 72 hours after last injection to treat BE, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same BE. Any bleed at different location: considered as separate BE, regardless of time from last injection. EP: sum of all intervals of time during which participants treated with BIVV001 according to study arms and treatment regimens. ABR: estimated by NB model with total number of treated BE during EP as response variable and log-transformed EP duration (years) as offset variable. Spontaneous: bleeding without contributing factor (definite trauma/antecedent strenuous activity). Traumatic: bleeding with known/believed reason.
Time Frame: Baseline up to Week 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
episodes per participant per year | 2.78 [1.39 to 5.58] | 2.32 [1.30 to 4.13]

6. Secondary Outcome: Annualized Bleeding Rate by Type of Bleed (Spontaneous, Traumatic and Unknown Type)
Description: ABR: annualized number of treated bleeding episodes per participant per year. ABR = number of all BE during EP/total number of days during EP*365.25. EP reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. Treated BE: episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one was considered 1st injection to treat new BE in same location. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection. Spontaneous bleeding: BE without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic bleeding: BE with known/believed reason for bleed.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population.
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
episodes per participant per year
  Spontaneous | 0.17 [0.08 to 0.38] | 0.14 [0.04 to 0.53]
  Traumatic | 0.28 [0.14 to 0.55] | 0.59 [0.31 to 1.14]
  Unknown type | 0.03 [0.00 to 0.20] | 0.59 [0.12 to 3.02]

7. Secondary Outcome: Sensitivity Analysis: Annualized Bleeding Rate by Type of Bleed (Spontaneous, Traumatic and Unknown Type)
Description: ABR: annualized number of treated bleeding episodes per participant per year. ABR = number of all BE during EP/total number of days during EP*365.25. EP reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. Treated BE: episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection. Spontaneous bleeding: BE without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic bleeding: BE with known/believed reason for bleed.
Time Frame: Baseline up to Week 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
episodes per participant per year
  Spontaneous | 0.17 [0.08 to 0.38] | 0.15 [0.04 to 0.55]
  Traumatic | 0.28 [0.14 to 0.55] | 0.52 [0.26 to 1.04]
  Unknown type | 0.03 [0.00 to 0.20] | 0.09 [0.03 to 0.27]

8. Secondary Outcome: Annualized Bleeding Rate by Location of Bleed (Joint, Muscle, Internal and Skin/Mucosa)
Description: ABR: annualized number of treated bleeding episodes per participant per year. ABR = number of all BE during EP/total number of days during EP*365.25. Efficacy period reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms and treatment regimens. Treated bleeding episode: episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection. Spontaneous bleeding: BE without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic bleeding: BE with known/believed reason for bleed.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
episodes per participant per year
  Joint | 0.19 (0.63) | 0.99 (3.62)
  Muscle | 0.03 (0.16) | 0.17 (0.51)
  Internal | 0.08 (0.28) | 0.06 (0.35)
  Skin/mucosa | 0.16 (0.38) | 0.25 (0.60)

9. Secondary Outcome: Sensitivity Analysis: Annualized Bleeding Rate by Location of Bleed (Joint, Muscle, Internal and Skin/Mucosa)
Description: ABR: annualized number of treated bleeding episodes per participant per year. ABR = number of all BE during EP/total number of days during EP*365.25. EP reflects sum of all intervals of time during which participants were treated with BIVV001 according to study arms & treatment regimens. Treated BE: episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode any subsequent bleeding at same location/injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection. Spontaneous bleeding: BE without contributing factor (definite trauma/antecedent "strenuous" activity). Traumatic bleeding: BE with known/believed reason for bleed.
Time Frame: Baseline up to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
episodes per participant per year
  Joint | 0.19 (0.63) | 0.40 (0.93)
  Muscle | 0.03 (0.16) | 0.17 (0.52)
  Internal | 0.08 (0.28) | 0.06 (0.35)
  Skin/mucosa | 0.16 (0.38) | 0.26 (0.61)

10. Secondary Outcome: Percentage of Participants Achieving FVIII Activity Levels Above 1%, 3%, 5%, 10%, 15%, and 20%
Description: FVIII activity level was measured using activated partial thromboplastin time (aPTT)-based one stage clotting assay. Percentage of participants who achieved steady-state trough FVIII activity levels above (>) 1%, 3%, 5%, 10%, 15%, and 20% were reported in this outcome measure. Participants were counted in more than one category, as applicable.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS. Here, 'overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 32 | 29
percentage of participants
  >1% | 100 | 100
  >3% | 100 | 100
  >5% | 75.0 | 100
  >10% | 18.8 | 51.7
  >15% | 9.4 | 6.9
  >20% | 3.1 | 6.9

11. Secondary Outcome: Number of Injections of BIVV001 Required to Treat a Bleeding Episode
Description: A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location was considered as separate bleeding episode, regardless of time from last injection.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS. Here, 'overall number of units analyzed' = total number of treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: injections per bleeding episode
Units Other Than Participants: Treated bleeding episode
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Number analyzed (Treated bleeding episode) | 17 | 47
injections per bleeding episode | 1.12 (0.33) | 1.30 (0.69)

12. Secondary Outcome: Sensitivity Analysis: Number of Injections of BIVV001 Required to Treat a Bleeding Episode
Description: A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS excluding 1 participant who did not receive weekly prophylaxis treatment as specified in the protocol for an extended period of time. Here, 'overall number of units analyzed' = total number of treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: injections per bleeding episode
Units Other Than Participants: Treated bleeding episode
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
Number analyzed (Treated bleeding episode) | 17 | 26
injections per bleeding episode | 1.12 (0.33) | 1.00 (0.00)

13. Secondary Outcome: Percentage of Bleeding Episodes Treated With a Single Injection of BIVV001
Description: A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection. Percentage of bleeding episodes (of all bleeding episodes occurred) which were treated with single injection was reported in this outcome measure.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population. Here, 'overall number of units analyzed' = total number of treated bleeding episodes.
Measure: Number; unit: percentage of bleeding episodes
Units Other Than Participants: Treated bleeding episode
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Number analyzed (Treated bleeding episode) | 17 | 47
percentage of bleeding episodes | 88.2 | 78.7

14. Secondary Outcome: Sensitivity Analysis: Percentage of Bleeding Episodes Treated With a Single Injection of BIVV001
Description: as for outcome 13
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS, excluding the participant who did not receive the weekly prophylaxis treatment as per protocol for an extended period of time. Here, 'overall number of units analyzed' = total number of treated bleeding episodes.
Measure: Number; unit: percentage of bleeding episodes
Units Other Than Participants: Treated bleeding episode
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
Number analyzed (Treated bleeding episode) | 17 | 26
percentage of bleeding episodes | 88.2 | 100

15. Secondary Outcome: Total Dose of BIVV001 Required to Treat a Bleeding Episode
Description: A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection. Total dose was expressed in unit: International units per kilogram (IU/kg).
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS. Here, 'overall number of units analyzed' = total number of treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Treated bleeding episode
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Number analyzed (Treated bleeding episode) | 17 | 47
IU/kg | 52.29 (15.84) | 66.90 (37.01)

16. Secondary Outcome: Sensitivity Analysis: Total Dose of BIVV001 Required to Treat a Bleeding Episode
Description: A bleeding episode was defined as an episode that started from 1st sign of bleed and ended no more than 72 hours after last injection to treat bleeding episode, any subsequent bleeding at same location or injections administered <=72 hours apart from previous injection were considered same bleeding episode. Any injection to treat bleed, taken >72 hours after preceding one, was considered 1st injection to treat new BE in same location. Any injection after >72 hours post preceding one, was considered 1st injection to treat new BE in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection. Total dose was expressed in unit: IU/kg.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS, excluding 1 participant who did not receive weekly prophylaxis treatment for an extended period of time. Here, 'overall number of units analyzed' = total number of treated bleeding episodes.
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Treated bleeding episode
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
Number analyzed (Treated bleeding episode) | 17 | 26
IU/kg | 52.29 (15.84) | 50.39 (6.71)

17. Secondary Outcome: Physicians' Global Assessment (PGA) of Participant's Response to BIVV001 Treatment Based on a 4-point Response Scale
Description: Physicians assessed participant's response to BIVV001 treatment using 4-point response scale categorized as: Excellent= BE responded to fewer than/usual number of injections/less than/usual dose of FVIII/rate of breakthrough bleeding during prophylaxis was <= that usually observed; Effective = most BE responded to same number of injections and dose, but some required more injections/higher doses/there was minor increase in rate of breakthrough bleeding; partially effective = BE most often required more injections and/or higher doses than expected/adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses; Ineffective = routine failure to control hemostasis or hemostatic control required additional agents.
Time Frame: Week 13 and Week 52/End of study (EOS)/Early termination (ET)
Population: Analysis was performed on FAS. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 37 | 36
Participants
  Week 13: Excellent | 37 | 34
  Week 13: Effective | 0 | 2
  Week 13: Partially effective | 0 | 0
  Week 13: Ineffective | 0 | 0
  Week 52/EOS/ET: Excellent | 37 | 36
  Week 52/EOS/ET: Effective | 0 | 0
  Week 52/EOS/ET: Partially effective | 0 | 0
  Week 52/EOS/ET: Ineffective | 0 | 0

18. Secondary Outcome: Participant's Response to BIVV001 Treatment Based on the International Society on Thrombosis and Haemostasis (ISTH) 4-point Response Scale
Description: Participant's response to the 1st injection of BIVV001 treatment for treating a bleed was evaluated by ISTH 4-point response scale categorized as: Excellent (complete pain relief/complete resolution of signs of bleeding), Good (significant pain relief /improvement in signs of bleeding), Moderate (modest pain relief/improvement in signs of bleeding) and none (no or minimal improvement/condition worsened). Assessed approximately 72 hours after initial treatment for BE. Bleeding episode: an episode that started from 1st sign of bleed and ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location/injections <=72 hours apart were considered same BE. Any injection after >72 hours post preceding one=considered 1st injection to treat new BE in same location. Any bleed at different location: considered as separate BE, regardless of time from last injection. Participants were counted in more than one category, as applicable.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population. Here, 'overall number of units analyzed' = number of injections with a response.
Measure: Count of Units; unit: Injections with a response
Units Other Than Participants: Injections with a response
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Number analyzed (Injections with a response) | 16 | 24
Injections with a response
  Excellent | 14 | 22
  Good | 1 | 2
  Moderate | 1 | 0
  None | 0 | 0

19. Secondary Outcome: Total Annualized BIVV001 Consumption Per Participant
Description: Total annualized BIVV001 consumption (in IU/kg) was calculated for each participant as: Total IU/kg of BIVV001 during EP divided by total number of days during EP*365.25. EP reflects the sum of all intervals of time during which participants were treated with BIVV001 according to the study arms and treatment regimens.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population.
Measure: Mean (Standard Deviation); unit: IU/kg per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
IU/kg per participant per year | 3115.57 (488.64) | 2884.67 (207.88)

20. Secondary Outcome: Annualized Joint Bleeding Rate (AJBR)
Description: AJBR: annualized number of joint bleeding/participant/year. ABR = number of treated joint BE during EP divided by total number of days during EP*365.25. Joint BE: unusual sensation in joint ('aura') along with 1) increasing swelling/warmth over skin, joint; 2) increasing pain or 3) progressive loss of range of motion/difficulty in using limb compared to Baseline. BE: episode started from 1st sign of bleed & ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location/injections <=72 hours apart considered same BE. Any injection after >72 hours post preceding one=1st injection to treat new BE in same location. Any bleed at different location=separate BE, regardless of time from last injection. EP: sum of all intervals of time during which participants treated with BIVV001 per study arms and treatment regimens. ABR:NB model with total number of treated BE during EP (response variable) & log-transformed EP duration (offset variable).
Time Frame: Baseline up to Week 52
Population: Analysis was performed on FAS population.
Measure: Mean (95% Confidence Interval); unit: joint BE per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
joint BE per participant per year | 0.19 [0.06 to 0.62] | 0.99 [0.38 to 2.60]

21. Secondary Outcome: Sensitivity Analysis: Annualized Joint Bleeding Rate (AJBR)
Description: AJBR: annualized number of joint bleeding/participant/year. ABR = number of treated joint BE during EP divided by total number of days during EP*365.25. Joint BE: unusual sensation in joint ('aura') along with 1) increasing swelling/warmth over skin, joint; 2) increasing pain or 3) progressive loss of range of motion/difficulty in using limb compared to Baseline. BE: episode started from 1st sign of bleed & ended no more than 72 hours after last treatment for bleed, within which any symptoms of bleeding at same location/injections <=72 hours apart considered same BE. Any injection after >72 hours post preceding one=1st injection to treat new BE in same location. Any bleed at different location=separate BE, regardless of time from last injection. EP: sum of all intervals of time during which participants treated with BIVV001 per study arms and treatment regimens. ABR: NB model with total number of treated BE during EP (response variable) & log-transformed EP duration (offset variable).
Time Frame: Baseline up to Week 52
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: joint BE per participant per year
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 35
joint BE per participant per year | 0.19 [0.06 to 0.62] | 0.41 [0.19 to 0.89]

22. Secondary Outcome: Change From Baseline in Hemophilia Joint Health Score Domain Score at Week 52
Description: HJHS is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. Following domains were assessed for elbows, knee and ankle joints: swelling (score 0 = no swelling to 3=severe), duration of swelling (score 0 = no swelling and 1 = >=6 months), muscle atrophy (score 0 = none to 2 = severe), crepitus on motion (score 0 = none to 2=severe), flexion loss (score 0 = <5' to 3 = >20'), extension loss (score 0 = <5' to 3 = >20'), joint pain (score 0 = no pain through active range of motion to 2 = pain through active range) and strength (score 0 = holds test position with maximum resistance to 4 = trace/no muscle contraction), for each item 0 = no damage and higher score = severe damage.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
score on a scale
  Swelling: number analyzed (Participants) | 19 | 35
  Swelling | 0.0 (0.0) | -0.1 (0.6)
  Duration Of Swelling: number analyzed (Participants) | 19 | 35
  Duration Of Swelling | 0.1 (0.2) | -0.0 (0.2)
  Muscle Atrophy: number analyzed (Participants) | 19 | 35
  Muscle Atrophy | 0.0 (0.0) | -0.1 (0.4)
  Crepitus On Motion: number analyzed (Participants) | 19 | 35
  Crepitus On Motion | 0.1 (0.2) | -0.1 (0.5)
  Flexion Loss: number analyzed (Participants) | 19 | 35
  Flexion Loss | -0.9 (4.1) | -0.1 (0.6)
  Extension Loss: number analyzed (Participants) | 19 | 35
  Extension Loss | -0.2 (1.0) | 0.2 (0.9)
  Joint Pain: number analyzed (Participants) | 19 | 35
  Joint Pain | 0.0 (0.0) | 0.0 (0.4)
  Strength: number analyzed (Participants) | 18 | 33
  Strength | 1.3 (10.0) | -0.8 (4.2)

23. Secondary Outcome: Change From Baseline in Hemophilia Quality of Life Questionnaire (Haemo-QoL) Kids Short Version Total Score at Week 52 for Children Participants (Aged 4 to 7 and 8 to <12 Years)
Description: Haemo-QoL kids short version: used to measure physical and emotional impacts on quality of life in children & adolescent with hemophilia. It was administered to children & their caregivers. Short version for children containing 16 items (4 to 7 years) and 35 items (8 to <12 years) were selected in this study. This version covers 9 dimensions relevant for children's HRQoL (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia & treatment). Items were rated along 5 response options: never, seldom, sometimes, often and always, higher scores=greater impairment. Raw score for each domain were transformed to scale ranged between 0 to 100, where lower score=better HRQoL. Haem- A-QoL total score=average of all domain scores and ranged from 0 to 100, where lower scores=better QoL.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field signifies that no participants were aged 8 to <12 years in arm "BIVV001: Participants aged <6 Years".
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 10 | 14
score on a scale
  4 to 7 years: number analyzed (Participants) | 10 | 4
  4 to 7 years | -5.31 (10.83) | 4.69 (5.41)
  8 to <12 years: number analyzed (Participants) | 0 | 10
  8 to <12 years |  | -9.79 (12.18)

24. Secondary Outcome: Change From Baseline in Hemophilia Quality of Life Questionnaire Parent Proxy Short Version Total Score at Week 52 for Children Participants (Aged 4 to 7 and 8 to <12 Years): Parent's Evaluation
Description: Haemo-QoL parent proxy short version: used to measure physical and emotional impacts on quality of life in children and adolescent with hemophilia. It was administered to children & their caregivers. Short version for children's caregivers containing 16 items (participants 4 to 7 years) and 35 items (participants 8 to <12 years) were selected in this study. This version covers 9 dimensions relevant for children's HRQoL (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia and treatment). Items are rated along 5 response options: never, seldom, sometimes, often and always, higher scores=greater impairment. Raw score for each domain: transformed to scale ranged between 0 to 100, lower score=better HRQoL. Haem-A-QoL total score=average of all domain scores and ranged from 0 to 100, lower scores=better quality of life. Haemo-QoL Total Score as per parent's evaluation was reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 19 | 13
score on a scale
  4 to 7 years: number analyzed (Participants) | 19 | 4
  4 to 7 years | -3.21 (12.23) | -1.17 (11.08)
  8 to <12 years: number analyzed (Participants) | 0 | 9
  8 to <12 years |  | -4.05 (10.77)

25. Secondary Outcome: Change From Baseline in Hemophilia Quality of Life Questionnaire Kids Short Version Physical Health Domain Score at Week 52 for Children Participants (Aged 8 to <12 Years)
Description: Haemo-QoL kids short version: used to measure physical and emotional impacts on quality of life in children and adolescent with hemophilia. It was administered to children and their caregivers. Short version for children containing 35 items (8 to <12 years) were selected in this study. This version covers 9 dimensions considered relevant for the children's HRQoL (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia and treatment). Items are rated along 5 response options: never, seldom, sometimes, often and always, higher scores=greater impairment. Raw score for physical health domain were transformed to scale ranged between 0 to 100, where lower score=better HRQoL. Change from baseline in physical Health domain score was reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS population. Here, 'Overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for arm 'BIVV001: Participants aged <6 years'.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 10
score on a scale | -10.63 (14.75)

26. Secondary Outcome: Change From Baseline in Hemophilia Quality of Life Questionnaire Parent Proxy Short Version Physical Health Domain Score at Week 52 for Children Participants (Aged 8 to <12 Years): Parent's Evaluation
Description: Haemo-QoL parent proxy short version: used to measure physical & emotional impacts on quality of life in children & adolescent with hemophilia. It was administered to children & their caregivers. Short version for children's caregivers containing 35 items (participants 8 to <12 years) were selected in this study. This version covers 9 dimensions relevant for children's HRQoL (physical health, feelings, view of yourself, family, friends, other people, sports and school, dealing with hemophilia & treatment). Items are rated along 5 response options: never, seldom, sometimes, often and always, higher scores=greater impairment. Raw score for physical health domain were transformed to scale ranged between 0 and 100, where lower score=better HRQoL. Change from baseline in physical health domain score as per parent's evaluation was reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 9
score on a scale | -7.64 (11.60)

27. Secondary Outcome: Total Number of Target Joints Resolved in Participants at Week 52
Description: A target joint at Baseline was defined as a major joint with >=3 spontaneous bleeding episodes in a consecutive 6 month period prior to entry to the study, captured at Baseline. A target joint resolved was defined as <=2 spontaneous bleeds into that joint during 12 months of continuous exposure (defined as treatment regimen period >=52 weeks). Total number of target joints resolved at Week 52 were reported.
Time Frame: Week 52
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and had at least 12 months of continuous exposure. 'Overall number of units analyzed' = total number of target joints at Baseline from participants with at least 12 months continuous exposure. Here "0" in 'overall number of participants analyzed' signifies that none of the participants had at least 12 months of continuous exposure.
Measure: Number; unit: Target joints resolved
Units Other Than Participants: Total number of target joints
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 0 | 1
Number analyzed (Total number of target joints) | 0 | 2
Target joints resolved |  | 2

28. Secondary Outcome: Change From Baseline in Hemophilia Joint Health Score (HJHS) Total Score at Week 52
Description: HJHS is a validated 11-item scoring tool developed for the assessment of joint health in participants with hemophilia. It comprised an evaluation of the elbows, knee and ankle joints: swelling (0 to 3), duration of swelling (0 to 1), muscle atrophy (0 to 2), crepitus on motion (0 to 2), flexion loss (0 to 3), extension loss (0 to 3), joint pain (0 to 2) and strength (0 to 4), in each item 0 = none and higher score = severe damage and global gait (walking, stairs, running, hopping on 1 leg) scored on scale ranged from 0 to 4, where 0 = all skills in normal limit and 4 = no skills within normal limits). Total HJHS score = sum of joint totals (0 to 120) + general gait (1 to 4) and ranged from 0 (no joint damage) to 124 (severe joint damage), where higher score indicated severe joint damage.
Time Frame: Baseline, Week 52
Population: Analysis was performed on FAS population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 18 | 33
score on a scale | 0.2 (8.3) | -1.1 (4.3)

29. Secondary Outcome: Investigators' or Surgeons' Assessment of Participant's Hemostatic Response to BIVV001 Treatment
Description: The Investigators/Surgeons who complete the surgical procedures assess the participant's response to surgery with BIVV001 treatment using a 4-point scale, where responses were categorized as: 1 = Excellent, 2 = Good, 3 = Fair, and 4 = Poor/none. Higher score indicated worst response. This assessment was performed 24 hours after the surgery. A surgery can be counted in more than one response category. As pre-specified, this outcome measure was planned to be analyzed combinedly for both the cohorts (participants <6 years and participants 6 to <12 years) and presented under a single reporting group.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on a surgery subgroup population which included all participants who had undergone major surgery after the 1st dose of study drug. Here, 'overall number of participants analyzed' = participants with major surgeries during the specified period (defined as the date and time of the first dose of study drug up to the last dose of study drug) and 'overall number of units analyzed' = number of major surgeries during the specified period occurred in participants analyzed.
Measure: Number; unit: major surgeries
Units Other Than Participants: Number of major surgeries
Groups:
- Participants With Major Surgery: Participants from any arm (BIVV001: participants aged <6 Years or BIVV001: participants aged 6 to <12 Years) who had at least 6 days of exposure to BIVV001 and a negative inhibitor test within 4 weeks prior to surgery and underwent major surgery (defined as any invasive operative procedure that required any of the following: opening into a major body cavity [e.g., abdomen, thorax, skull]; operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier [e.g., pleura, peritoneum, dura]) after the first dose of study drug during the study.
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgeries) | 2
major surgeries
  Excellent or Good | 2
  Excellent | 2
  Good | 0
  Fair | 0
  Poor/none | 0

30. Secondary Outcome: Number of Injections Per Surgery Required to Maintain Hemostasis During Perioperative Period for Major Surgery
Description: Perioperative period was time lapse surrounding the surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). The number of injections to maintain hemostasis (process to prevent and stop bleeding from blood vessel) per surgery included all injections from loading dose (i.e., the preoperative injection, administered either on the day of surgery or one day prior to the surgery), to end of surgery. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: During the perioperative period (any time during Baseline up to Week 52)
Population: Analysis was performed on surgery subgroup population. Here, 'overall number of participants analyzed' = participants with major surgeries during the specified period and 'overall number of units analyzed' = number of major surgeries during the specified period occurred in participants analyzed. As pre-specified, this outcome measure was planned to be analyzed combinedly for both the cohorts (participants <6 years and participants 6 to <12 years) and presented under a single reporting group.
Measure: Number; unit: Major surgeries
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgeries) | 2
Major surgeries
  One injection | 2
  Two injection | 0
  Three injection | 0
  Four injection | 0
  >Four injection | 0

31. Secondary Outcome: Number of Blood Component Transfusions Used During Perioperative Period for Major Surgery
Description: The perioperative period was the time lapse surrounding the surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). The number of blood component transfusions used during perioperative period were summarized categorically (0, 1, 2, 3 and >3) for all major surgeries for the surgery subgroup. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: During the perioperative period (any time during Baseline up to Week 52)
Population: as for outcome 30
Measure: Number; unit: Major surgeries
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgeries) | 2
Major surgeries
  Zero | 2
  One | 0
  Two | 0
  Three | 0
  >Three | 0

32. Secondary Outcome: Total BIVV001 Consumption From Day -1 to 14 During Perioperative Period for Major Surgery
Description: Perioperative period: time lapse surrounding surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). Total BIVV001 consumption were summarized from the loading dose (the day before surgery, i.e., on Day -1) up to 2 weeks following the surgery (i.e., Day 14) and were reported in this outcome measure.
Time Frame: Day -1 to Day 14
Population: Analysis was performed on surgery subgroup population. Here, 'overall number of participants analyzed' = participants with major surgeries during the specified period and 'overall number of units analyzed' = number of major surgeries with BIVV001 administration within Day -1 to Day 14. As pre-specified, this outcome measure was planned to be analyzed combinedly for both the cohorts (participants <6 years and participants 6 to <12 years) and presented under a single reporting group.
Measure: Mean (Standard Deviation); unit: IU/kg per major surgery
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgeries) | 2
IU/kg per major surgery | 201.97 (29.42)

33. Secondary Outcome: Type of Blood Component Transfusions Used During Perioperative Period for Major Surgery
Description: The perioperative period was the time lapse surrounding the surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during the surgery) and post-operative (24-hour post-surgery). The type of blood component (Red blood cell, platelet, fresh frozen plasma, whole blood and other) transfusions used were summarized for all major surgeries. Post-operative referred to the day following the end of surgery to the date of hospital discharge. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: During the perioperative period (any time during Baseline up to Week 52)
Population: as for outcome 30
Measure: Number; unit: Major surgeries
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgeries) | 2
Major surgeries
  Red Blood Cell | 0
  Platelet | 0
  Fresh Frozen Plasma | 0
  Whole Blood | 0
  Other | 0

34. Secondary Outcome: Total Dose Required to Maintain Hemostasis From Day -1 to Day 0 During Perioperative Period for Major Surgery
Description: Perioperative period was time lapse surrounding surgical act which was divided into 3 stages: preoperative (4 weeks prior to surgery), operative (during surgery) and post-operative (24-hour post-surgery). Total dose (IU/kg) was sum across all injections per major surgery (including loading dose) needed to maintain hemostasis (process to prevent and stop bleeding from blood vessel) during surgery. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on joint; removal of organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of mesenchymal barrier (e.g., pleura, peritoneum, dura). Day 0=surgery day. Loading dose for given surgery was preoperative injection, administered either on day of surgery or one day prior to surgery (i.e., Day -1).
Time Frame: Day -1 to Day 0 (day of surgery)
Population: Analysis was performed on surgery subgroup population. Here, 'overall number of participants analyzed' = participants with major surgeries during the specified period and 'overall number of units analyzed' = number of major surgeries for which a loading dose was given on the day of surgery or one day prior to surgery (i.e. Day -1). As pre-specified, this outcome measure was planned to be analyzed combinedly for both the cohorts and presented under a single reporting group.
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Number of major surgeries
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgeries) | 2
IU/kg | 61.13 (1.06)

35. Secondary Outcome: Estimated Blood Loss During Major Surgery
Description: The estimated total blood loss (in milliliters) during major surgeries were summarized. Major surgery: defined as any invasive operative procedure that required any of the following: opening into major body cavity (e.g., abdomen, thorax, skull); operation on a joint; removal of an organ; dental extraction of any molar teeth or >=3 non-molar teeth; operative alteration of normal anatomy; crossing of a mesenchymal barrier (e.g., pleura, peritoneum, dura).
Time Frame: Day 0 (i.e., day of surgery)
Population: Analysis was performed on surgery subgroup population. Here, 'overall number of participants analyzed' = participants with reported blood loss during major surgery and 'overall number of units analyzed' = number of major surgeries with blood loss report during the treatment regimen occurred in participants analyzed. As pre-specified, this outcome measure was planned to be analyzed combinedly for both the cohorts and presented under a single reporting group.
Measure: Mean (Standard Deviation); unit: milliliters
Units Other Than Participants: Number of major surgery with blood loss
Arm/Group | Participants With Major Surgery
Number analyzed (Participants) | 2
Number analyzed (Number of major surgery with blood loss) | 2
milliliters | 25.00 (35.36)

36. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug which did not necessarily have a causal relationship with the treatment. A serious AE (SAE) was defined as any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly or birth defect, or was a medically important event. Treatment-emergent AEs were AEs that developed, worsened or became serious from Baseline (Day 1) up to 3 weeks post last dose.
Time Frame: From Baseline (Day 1) up to 3 weeks post last dose of BIVV001 (i.e., up to Week 55)
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Participants
  TEAE | 33 | 29
  TESAE | 5 | 4

37. Secondary Outcome: Number of Participants With Occurrence of Embolic and Thrombotic Events
Description: Embolic and thrombotic events were defined as arterial or venous thrombosis, confirmed by imaging.
Time Frame: Baseline up to Week 52
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
Number analyzed (Participants) | 38 | 36
Participants | 0 | 0

38. Secondary Outcome: Pharmacokinetics (PK): Maximum FVIII Activity (Cmax)
Description: Cmax was defined as the maximum observed plasma FVIII Activity.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: Analysis was performed on PK population which included all participants who had completed adequate blood sample collection to assess key PK parameters. Data was planned to be collected and analyzed for combined population of both arm groups with the available PK data.
Measure: Mean (Standard Deviation); unit: IU per decilitre
Groups:
- BIVV001 (Efanesoctocog Alfa): All participants who were enrolled in study and received BIVV001 in either Arm 'BIVV001: participants aged <6 years' or 'BIVV001: participants aged 6 to <12 years'.
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 37
IU per decilitre | 128 (46.4)

39. Secondary Outcome: Pharmacokinetics: Clearance (CL)
Description: CL is defined as the rate at which the drug is removed from the body.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: Analysis was performed on PK analysis set. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data was planned to be collected and analyzed for combined population of both arm groups with the available PK data.
Measure: Mean (Standard Deviation); unit: millilitres per hour per kilogram
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 36
millilitres per hour per kilogram | 0.711 (0.132)

40. Secondary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution (Vd) is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: milliliters per kilogram
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 36
milliliters per kilogram | 37.3 (6.19)

41. Secondary Outcome: Pharmacokinetics: Elimination Half-life (t1/2z)
Description: Plasma t1/2z was the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 36
hours | 40.2 (4.29)

42. Secondary Outcome: Pharmacokinetics: Area Under the Plasma FVIII Activity Versus Time Curve (AUC0-tau)
Description: AUC0-tau was defined as area under the plasma concentration-time profile from time zero (pre-dose) to dosing interval.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: hour*IU per deciliter
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 35
hour*IU per deciliter | 7000 (1300)

43. Secondary Outcome: Pharmacokinetics: Total Clearance at Steady State (CLss)
Description: CLss is defined as the rate at which the drug is removed from the body at steady state.
Time Frame: 0 hour - 168 hour at week 26, 39 or 52
Population: Data for this outcome measure is not reported because samples were not collected to estimate CLss.
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 0

44. Secondary Outcome: Pharmacokinetics: Incremental Recovery (IR)
Description: IR was calculated as (Peak activity [in IU/dL] - Trough activity [in IU/dL])/Actual Dose (in IU/kg), and peak activity at each visit was the highest activity level after the dosing, and trough activity at each visit was the activity level prior to the dosing.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: Analysis was performed on PK analysis set. Data was planned to be collected and analyzed for combined population of both arm groups with the available PK data.
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 37
IU/dL per IU/kg | 2.53 (0.880)

45. Secondary Outcome: Pharmacokinetics: Trough Concentration for BIVV001 (Ctrough)
Description: Ctrough is the pre-dose concentration of a drug. Ctrough was measured by apTT-Baseline-one-stage clotting assay.
Time Frame: Pre-dose at Baseline (Day 1) and Week 52
Population: Analysis was performed on FAS population. Here, 'number analyzed' = participants with available data for each specified category. Data was planned to be collected and analyzed for combined population of both arm groups with the available PK data.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 74
IU/dL
  Baseline: number analyzed (Participants) | 69
  Baseline | 0.00 (0.00)
  Week 52: number analyzed (Participants) | 72
  Week 52 | 13.68 (21.84)

46. Secondary Outcome: Pharmacokinetics: Mean Residence Time (MRT)
Description: MRT is the average total time a drug molecule spends in the body.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 36
hours | 53.0 (6.22)

47. Secondary Outcome: Time Above Predefined (10% and 40%) FVIII Activity Levels
Description: Time above predefined (10% and 40%) FVIII activity levels mean time which BIVV001 maintains above 10 IU/dL and 40 IU/dL with single doses of 50 IU/kg.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: Analysis was performed on PK analysis set. Here, 'number analyzed' = participants with available data for each specified category. Data was planned to be collected and analyzed for combined population of both arm groups with the available PK data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 37
hours
  Time to 10 IU/dL | 160 (18.7)
  Time to 40 IU/dL | 72.2 (12.5)

48. Secondary Outcome: Pharmacokinetics: Dose-normalized Area Under the Activity-time Curve (DNAUC0-tau)
Description: AUC0-tau was defined as the area under the activity-time curve over the dosing interval. AUC was normalized by dose.
Time Frame: Pre-dose, 0.25, 3, 24, 72, and 168 hours post-dose on Day 1
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: hour*kilogram*IU/deciliter/IU
Arm/Group | BIVV001 (Efanesoctocog Alfa)
Number analyzed (Participants) | 35
hour*kilogram*IU/deciliter/IU | 139 (25.2)

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) up to 3 weeks post last dose of BIVV001 (i.e., up to Week 55)
Description: Analysis was performed on safety analysis set.
Arm/Group | BIVV001: Participants Aged <6 Years | BIVV001: Participants Aged 6 to <12 Years
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 5/38 | 4/36
Other Adverse Events (participants affected / at risk) | 31/38 | 28/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIVV001: Participants Aged <6 Years (N=38) | BIVV001: Participants Aged 6 to <12 Years (N=36)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Vascular Device Infection (Infections and infestations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vascular Device Occlusion (General disorders) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Circumcision (Surgical and medical procedures) | 1 (1) | 0 (0)
Device Malfunction (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIVV001: Participants Aged <6 Years (N=38) | BIVV001: Participants Aged 6 to <12 Years (N=36)
Asymptomatic Covid-19 (Infections and infestations) | 2 (2) | 5 (5)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2)
Ear Infection (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 5 (6) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (6) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory Tract Infection Viral (Infections and infestations) | 2 (3) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 5 (7)
Viral Infection (Infections and infestations) | 3 (4) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 (4) | 1 (2)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Peripheral Swelling (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (17) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0)
Sars-Cov-2 Test Positive (Investigations) | 7 (7) | 4 (6)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04759131/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04759131/SAP_001.pdf